CLINICAL TRIAL: NCT06968351
Title: Animal-Assisted Intervention: An Effectiveness Study Using Qualitative and Quantitative Measures on Offenders With Mental Illnesses in Hong Kong
Brief Title: A Pilot Study on Animal-Assisted Intervention in Correctional Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Correctional Services Department (Unknown)
Responsible Party: Principal Investigator, Amanda Kingsze CHEUNG, Research Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA240679
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Psychological Wellbeing; Animal-assisted Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants are assigned to a brief animal-assisted intervention that is offered on a group basis across four sessions. Each of the four sessions lasts approximately 60 minutes. In addition to questionnaire data prior to and after the treatment, participants will provide physiological and questionnaire data at both the beginning and the end of each session.
  Interventions: Behavioral: Animal-Assisted Intervention

INTERVENTIONS:
Behavioral: Animal-Assisted Intervention — A brief animal-assisted intervention is offered on a group basis across four sessions. Each session lasts approximately 60 minutes and covers the same themes but through different exercises. These themes include effective communication, behavioral principles, problem-solving, and teamwork. The first part of a session involves learning to give effective single-component commands to a rehabilitative dog under the guidance of a professional dog handler. The second part of a session involves the applications of two or more of these single-component commands to an interactive group activity. Project staff are present at each session to facilitate discussions among participants on any challenges encountered, learning, and intra- as well as inter-personal experiences during the session.
  Other Names: AAI; Dog Therapy

SUMMARY:
Mental health concerns such as depression, anxiety, and post-traumatic stress are particularly prevalent among incarcerated individuals and are considered risk factors for recidivism. Leveraging the natural human-animal bond, animal-assisted intervention (AAI) offers a less threatening alternative to engage incarcerated individuals and address their mental health needs. As an initial effort to help promote rehabilitative security in Hong Kong, the current study examines the acceptability and effectiveness of a brief animal-assisted program among offenders in local secured facilities.

ELIGIBILITY:
Inclusion Criteria:

* persons-in-custody
* aged 18 or older
* understand Cantonese

Exclusion Criteria:

* an allergy, a fear, or a dislike toward dogs
* a history of aggression toward animals
* a criminal history involving animals
* a history of neurodevelopmental disorders
* active psychosis or mania
* active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in common psychopathology as measured with the Depression, Anxiety, and Stress Scale - 21 Items | At the beginning of each sessions, approximately one week after completion of the treatment, and one month after the treatment
  Depression, Anxiety, and Stress Scale - 21 Items (DASS21; Lovibond & Lovibond, 1995) is a self-report measure of common mental health concerns. The three subscales are each measured with seven items, using a 4-point Likert scale from 0 = Did not apply to me at all to 3 = Applied to me very much or most of the time. Scores are summed for each subscale, with higher scores indicating more severe levels of emotional symptoms.
Change in emotional state as measured with the International Positive and Negative Affect Schedule Short Form | At the beginning and at the end of each session, up to a total of four sessions
  International Positive and Negative Affect Schedule Short Form (I-PANAS-SF; Thompson, 2007) is an adapted version of the PANAS-SF (Watson et al., 1988) and designed specifically for non-English speaking individuals. Using a 5-point Likert scale from 1 = Never to 5 = Always, individuals rate on their experience of five positive affect and five negative affect in the present moment. Scores are summed for each subscale, with higher scores indicating higher levels of positive or negative affect.
Change in heart rate variability | At the beginning and at the end of each session, up to a total of four sessions
  Heart rate data are collected via photoplethysmogram signals and then transformed into heart rate variability with artifacts corrected through automated detection using the Kubios HRV Scientific software (Kubios, 2024).
Change in skin conductance | At the beginning and at the end of each session, up to a total of four sessions
  Both phasic and tonic skin conductance data are captured with a galvanic skin response sensor

SECONDARY OUTCOMES:
Change in disciplinary offences and privileges during incarceration | At each session, up to a total of four sessions, and within a week after the treatment
  To track PIC's conduct and interpersonal behaviors during incarceration, official correctional records on disciplinary offences and privileges received in the week prior to each AAI session, including counts and associated behaviors, are collected.
Change in trauma-related psychopathology as measured with the Posttraumatic Stress Disorder Checklist for DSM-5 | Before treatment, within a week after treatment, and one month after treatment
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a self-report measure of posttraumatic stress disorder (PTSD) symptom severity, based on its diagnostic criteria in DSM-5 (Blevins et al., 2015). Each of the 20 items is rated on a 5-point Likert scale of 0 = Not at all to 4 = Extremely.
Change in empathy as measured with the Brief Interpersonal Reactivity Index | Before treatment, within a week after treatment, and one month after treatment
  Brief Interpersonal Reactivity Index (B-IRI) measures empathy by four subscales, namely Perspective Taking, Empathic Concern, Fantasy, and Personal Distress. Each subscale is measured by four items, using a 5-point Likert scale from 1 = Does not describe me at all to 5 = Describes me very well and with higher sum scores indicating higher levels in the corresponding aspect of empathy.
Change in self-efficacy as measured with the New General Self-Efficacy Scale | Before treatment, within a week after treatment, and one month after treatment
  New General Self-Efficacy Scale (NGSES) is designed to measure self-efficacy across contexts. Using a 5-point Likert scale from 1 = Strongly disagree to 5 = Strongly agree, individuals rate on a total of eight items about their self-perceived ability to perform across different contexts. Scores are summed across all items, with higher scores indicating greater self-efficacy.
Change in psychological flexibility as measured with the Multidimensional Psychological Flexibility Inventory | Before treatment, within a week after treatment, and one month after treatment
  The Multidimensional Psychological Flexibility Inventory (MPFI; Rolffs et al., 2018) measures an individual's flexibility in responding to difficult experiences. Its short form consists of 12 items, which uses a 6-point Likert scale from 1 = Never True to 6 = Always True, and demonstrates psychometric soundness when used among Chinese (Li, 2024). Scores are summed across items, with higher scores indicate greater level of psychological flexibility.
Change in openness to treatment as measured with the Attitudes Toward Seeking Professional Psychological Help | Before treatment, within a week after treatment, and one month after treatment if feasible
  Attitudes Toward Seeking Professional Psychological Help (ATSPPH) measures an individual's help seeking preferences as indicated by three subscales, namely Openness to seeking professional help, Value in seeking professional help, and Preference to cope on one's own. Its short form contains 10 items, each rated on a 4-point Likert scale from 0 = Disagree to 3 = Agree. Scores are summed across items for each subscale, with higher scores indicating greater levels in each of the measured domains.
Change in social interactions | At each session, up to a total of four sessions, and within a week after the treatment
  Participants' behaviors during each AAI session and across the sessions are rated by independent observers on six items, using 3- to 5-point Likert scales (Koda et al., 2015). These items ask for ratings on a participant's general facial expression in terms of its affective valence, tenderness toward the animal, amount of talking, willingness to have contact with the animal, interest in the animal, and ease of interaction with the animal.
Subjective experience with the treatment | Within a month after the treatment
  Four open-ended questions are used to help understand participants' experience with the AAI descriptively. These items include one on overall psychological wellbeing on the day of measurement, one on feelings toward the animal, one on feelings toward peers in the assigned AAI, and one on overall psychological wellbeing throughout the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Correctional Services Department, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Sensitive data are collected and no authorization is obtained from study participants.